CLINICAL TRIAL: NCT04133948
Title: Multicenter Phase 1b Trial Testing the Neoadjuvant Combination of Domatinostat, Nivolumab and Ipilimumab in IFN-gamma Signature-low and IFN-gamma Signature-high RECIST 1.1-measurable Stage III Cutaneous or Unknown Primary Melanoma
Acronym: DONIMI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: 4SC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M19DON
Record Dates: First submitted 2019-10-14; First posted 2019-10-21 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Malignant Melanoma Stage III
Keywords: Melanoma; Neo-adjuvant; Domatinostat; Nivolumab; Ipilimumab
MeSH Terms: conditions — Melanoma | interventions — domatinostat; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A (Experimental): For IFN-gamma high patients: patients will receive pre-surgically 2 courses nivolumab 240 mg (q3weeks)
  Interventions: Drug: Nivolumab
- B (Experimental): For IFN-gamma high patients: patients will receive pre-surgically 2 courses nivolumab 240 mg (q3weeks) + domatinostat 200 mg BID, on days 1-14 (q3weeks)
  Interventions: Drug: Domatinostat; Drug: Nivolumab
- C (Experimental): For IFN-gamma low patients: patients will receive pre-surgically 2 courses nivolumab 240 mg (q3weeks) + domatinostat 200 mg BID, on days 1-14 (q3weeks)
  Interventions: Drug: Domatinostat; Drug: Nivolumab
- D (Experimental): For IFN-gamma low patients: patients will receive pre-surgically 2 courses nivolumab 240 mg (q3weeks) + ipilimumab 80 mg (q3weeks) + domatinostat. Patients in arm D will start with once daily (OD) dosing scheme of domatinostat 200 mg, on days 1-14 (q3weeks). Based on safety data of the first 5 patients in this arm, the next patients will be treated with either a higher dosing scheme (200 mg BID, days 1-14, q3weeks), a lower dosing scheme (100 mg OD, days 1-14, q3weeks), or the same dosing scheme (200 mg OD, days 1-14, q3weeks).
  Interventions: Drug: Domatinostat; Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Domatinostat — Patients in arm B and C will receive domatinostat 200 mg BID, days 1-14 q3weeks.
  Patients in arm D will start with once daily (OD) dosing scheme of domatinostat 200mg, d1-14 q3wks. Based on safety data of the first 5 patients in this arm, the next patients will be treated with either a higher dosing scheme (200mg BID, d1-14, q3wks), a lower dosing scheme (100mg OD, d1-14, q3wks) or the same dosing scheme (200mg OD, d1-14, q3wks).
  Arms: B; C; D
Drug: Nivolumab — 2 courses nivolumab 240 mg q3weeks
Drug: Ipilimumab — 2 courses ipilimumab 80 mg q3weeks
  Arms: D

SUMMARY:
DONIMI is a phase 1b trial testing the combination of domatinostat + nivolumab or nivolumab monotherapy in IFN-gamma signature high patients and of domatinostat + nivolumab or domatinostat + nivolumab + ipilimumab in IFN-gamma signature low patients with de-novo or recurrent macroscopic stage III cutaneous or unknown primary melanoma.

The trial will include 45 stage III cutaneous or unknown primary melanoma patients with RECIST 1.1 measurable de-novo or recurrent disease (short axis lymph node metastasis ≥1.5cm).

NanoString IFN-gamma signature high patients will be randomized to be treated pre-surgically for 6 weeks with nivolumab (arm A; 10 patients) or domatinostat + nivolumab (arm B; 10 patients).

IFN-gamma signature low patients will be randomized to be treated pre-surgically for 6 weeks with domatinostat + nivolumab (arm C; 10 patients) or domatinostat + nivolumab + ipilimumab (arm D; 15 patients). Patients will be stratified according to center.

Post-surgery (starting at week 12), the patients will start with adjuvant nivolumab or pembrolizumab for 52 weeks according to institute's standard. BRAF V600E/K mutation positive patients with no pathologic response after neoadjuvant therapy may also receive adjuvant BRAF + MEK inhibition if commercially available and according to the patient's and the treating physician's decision.

Follow-up after the adjuvant therapy will be for 2 years, according to the institutes' standard.

Toxicity and pathologic response rates will be descriptive. In case of 2/5 or 4/10 patients not undergoing their lymph node dissection at week 6 +/- 1 week due to treatment related toxicity, this arm will be declared unfeasible.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age.
* World Health Organization (WHO) Performance Status 0 or 1.
* Cytologically or histologically confirmed resectable stage III cutaneous melanoma (unknown primary also allowed) with one or more macroscopic lymph node metastases (measurable according to RECIST 1.1), that can be biopsied, and no history of in-transit metastases within the last 6 months.
* No other malignancies, except adequately treated and a cancer-related life-expectancy of more than 5 years.
* Patient willing to undergo quadruple tumor biopsies and extra blood withdrawal during screening, week 3 and in case of relapse.
* The biopsies at screening should contain at least 30% tumor cells in order to get a reliable IFN-gamma signature
* No immunosuppressive medications within 6 months prior trial registration.
* Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥1.5x109/L, Platelets ≥100 x109/L, Hemoglobin ≥5.5 mmol/L, Creatinine ≤1.5x ULN, AST ≤ 1.5 x ULN, ALT ≤ 1.5 x ULN, Bilirubin ≤1.5 X ULN.
* Normal LDH.
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of ipilimumab + nivolumab.
* Patient is capable of understanding and complying with the protocol requirements and has signed the Informed Consent document.

Exclusion Criteria:

Distantly metastasized melanoma

* Uveal or mucosal melanoma.
* History of in-transit metastases within the last 6 months.
* No measurable lymph node lesion according to RECIST 1.1.
* Subjects with any active autoimmune disease or a documented history of autoimmune disease, or history of syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy.
* Patients with any active gastrointestinal disorder that could interfere with the absorption of domatinostat (as per judgement of the investigator), such as ulcerative colitis, Crohn's disease, diabetic gastroparesis, or other syndromes characterized by malabsorption.
* Prior CTLA-4 or PD-1/PD-L1 targeting immunotherapy.
* Prior targeted therapy targeting BRAF and/or MEK.
* Prior radiotherapy.
* Patients will be excluded if they test positive for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody), indicating acute or chronic infection; if treated and being at least one year free from HCV patients are allowed to participate.
* Patients will be excluded if they have known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Allergies and Adverse Drug Reaction:

  * History of allergy to study drug components;
  * History of severe hypersensitivity reaction to any monoclonal antibody.
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity or adverse events.
* Patients with a marked baseline prolongation of QT/QTc interval, e.g., repeated demonstration of a QTc interval >450 msec (Grade 1 NCI-CTCAE); Long-QT-Syndrome) and patients receiving agents known to prolong the QT interval and known risk of Torsades de Pointes.
* Patients with significant current cardiovascular disease including:

  * Unstable angina pectoris within 6 months prior to screening
  * Uncontrolled hypertension
  * Congestive heart failure (New York Heart Association (NYHA) Class III or IV) related to primary cardiac disease
  * Conditions requiring anti-arrhythmic therapy (patients with status post pace maker implantation can be included)
  * Symptomatic ischemic or severe valvular heart disease, or a myocardial infarction within 6 months prior to the trial entry
* Women who are pregnant or lactating
* Use of other investigational drugs before study drug administration 30 days and 5 half-times before trial registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2022-01-11 (Actual); Study Completion 2024-11-26 (Actual)

PRIMARY OUTCOMES:
Safety of patients as measured by the adherence to the timelines in the study protocol | 6 months
  A treatment arm will be declared as not safe if 8/10 patients develop gr 3-4 adverse events or if 2/10 patients develop longlasting (>6 months) gr 3-4 adverse events.
Feasability of patients as measured by the adherence to the timelines in the study protocol | 6 weeks
  A treatment arm will be declared as not feasible if 2/5 or 4/10 patients cannot adhere to the planned time of surgery (week 6 +/- 1 week) due to treatment related adverse events.

SECONDARY OUTCOMES:
Pathologic response rates (pPR, near-pCR, and pCR). | At 6 weeks
Frequency of treatment-related toxicities as measured according to CTCAE 5.0. | At 6 weeks
Radiologic response rate according to RECIST 1.1 criteria | At 6 weeks
Relapse Free Survival (RFS) | Up to 3 years after treatment
RNA signatures associated with pathologic response and RFS for each arm (by RNAseq and NanoString gene expression analysis). | Up to 3 years after treatment
Changes in immune infiltrates/markers at week 3 and/or 6 compared to baseline by NanoString DSP technology or alternative immunohistochemistry analysis. | At week 3 and/or 6
Inter-arm comparison of the expansion of tumor-resident T cell clones, as measured by TCR sequencing of the baseline tumor-biopsy and PBMC samples from baseline week 3 and week 6. | At week 3 and/or 6
Feces microbiome diversity analyses and its correlation with pathologic response and toxicities. | Up to 3 years after treatment
Quality of life as measured by EORTC QLQ C30 | Up to 3 years after treatment
Quality of life as measured by the the Melanoma Subscale and Melanoma Surgery Subscale of FACT-M | Up to 3 years after treatment
Quality of life as measured by the Cancer Worry Scale | Up to 3 years after treatment
Quality of life as measured by HADS questionnaire | Up to 3 years after treatment
Quality of life as measured by EQ-5D-5L | Up to 3 years after treatment
Quality of life as measured by the immunotherapy-specific questionnaire | Up to 3 years after treatment
Quality of life as measured by an assessment of work performance. | Up to 3 years after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Christian Blank, Prof., Study Chair — Medical oncologist/researcher
Locations (2):
- Melanoma Institute Australia, Sydney, Wollstonecraft NSW, Australia
- Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215